CLINICAL TRIAL: NCT05766345
Title: BCG-induced Epigenetic Modifications in the NEXT Generation
Acronym: NEXT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 114192; 2023-503344-14-00 (Other: CTIS number (EMA))
Record Dates: First submitted 2023-01-16; First posted 2023-03-13 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-02

CONDITIONS: Trained Immunity; BCG Vaccine; Epigenetics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG vaccine (Experimental): BCG-Vaccine SSI [Statens Serum Institut]) Danish strain 1331 0.1ml (=0.0075mg) One-time vaccination intradermally
  Interventions: Biological: BCG-Vaccine SSI [Statens Serum Institut]) Danish strain 1331
- Placebo vaccine (Placebo Comparator): 0.9% NaCl placebo 0.1ml One-time vaccination intradermally
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: BCG-Vaccine SSI [Statens Serum Institut]) Danish strain 1331 — Nothing to add
  Arms: BCG vaccine
Biological: Placebo — Nothing to add
  Arms: Placebo vaccine

SUMMARY:
Non-specific protective effects resulting from the BCG vaccine appear to be paternally inheritable. Since the BCG vaccine is known to induce trained immunity, epigenetics might explain the fathers' contribution to the immune profile of their offspring. Epigenetic inheritance in mice has recently been demonstrated, but is not established in humans yet. By studying the DNA methylation profile of sperm cells after BCG vaccination, we aim to gain insight into the possibility of epigenetic inheritance in human males.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* Age 18-25 years (at the moment of trial start)

Exclusion Criteria:

* Any systemic disease or conditin, or the use of systemic medication (with the exception of non-threatening alelrgies, e.g. hay fever)
* Smoking or drug use
* Prior BCG vaccination
* Other vaccination four weeks prior to trial start or four weeks after the first study visit (no vaccine in the same arm as the BCG vaccine for three months)
* Acute illness two weeks prior to trial start
* Known allergy or history of anaphylaxis/other serious adverse reaction to any vaccine
* Participation in another drug trial
* Legally incapacitated or unwilling to provide informed consent

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The purpose of this study is to study sperm cells, therefore only male individuals can participate
Enrollment: 36 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
DNA methylation profile of sperm cells (first comparison; CHANGE) | Comparing T3 to baseline
  Differentially methylated regions (DMRs)
DNA methylation profile of sperm cells (second comparison; CHANGE) | Comparing T4 to baseline
  Differentially methylated regions (DMRs)

SECONDARY OUTCOMES:
Immunological profile of PBMCs, before and after BCG vaccination (comparison; CHANGE) | Comparing T1-T4 to baseline
  Cytokine production assays (e.g. TNFa, IL6, IL1b)
CHANGE of the epigenetic profile of innate immune cells | Comparing T1-T4 to baseline
  Differentially methylated regions (DMRs), ATAC sequencing, RNA sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No